CLINICAL TRIAL: NCT06927011
Title: Chronic Loose Stools Following Right-sided Hemicolectomy for Colon Cancer and the Association With Bile Acid Malabsorption and Small Intestinal Bacterial Overgrowth Using a Novel Sampling Device
Status: Not yet recruiting | Type: Observational
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 2024-0532; NCI-2025-02650 (Other: NCI-CTRP CLINICAL REGISTRY)
Record Dates: First submitted 2025-04-08; First posted 2025-04-15 (Actual); Last update posted 2025-10-23 (Actual); Status verified 2025-10

CONDITIONS: Colon Cancer
MeSH Terms: conditions — Colonic Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Colon Cancer: Participants will be asked to swallow 2 small devices (called Capscan), which will collect samples of intestinal fluid as they move through participants small intestine and colon. This device is not FDA approved but has been deemed to have no significant risk. The investigator can explain how it is designed to work. Participants will also answer surveys about participants quality of life.
  Participants in this study will be over after all study procedures are completed.
  Interventions: Behavioral: Capscan

INTERVENTIONS:
Behavioral: Capscan — Participants will be asked to swallow 2 small devices (called Capscan), which will collect samples of intestinal fluid as they move through participants small intestine and colon. This device is not FDA approved but has been deemed to have no significant risk. The investigator can explain how it is designed to work. Participants will also answer surveys about participants quality of life.
  Participants in this study will be over after all study procedures are completed.

SUMMARY:
The goal of this clinical research study is to learn about gastrointestinal symptoms in participants who have undergone SC or RC and their impact on the quality of life of these participants.

DETAILED DESCRIPTION:
To estimate the microbiota and bile acid profiles at multiple levels of the small intestine and proximal neo-colon in patients after RC and participants after SC.

ELIGIBILITY:
Inclusion Criteria:

* Both men and women of all races and ethnic groups are eligible for this trial who meet the above criteria.

Exclusion Criteria:

* Children will not be enrolled in this study.
* Pregnant women will not be enrolled in this study.
* Cognitively impaired subjects will not be enrolled in this study.

Ages: 20 Years to 85 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: MD Anderson Cancer Center
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2025-10-31 (Estimated); Primary Completion 2026-12-30 (Estimated); Study Completion 2028-12-30 (Estimated)

PRIMARY OUTCOMES:
Overall Survival (OS) | Through study completion; an average of 1 year.

CONTACTS AND LOCATIONS:
Locations (1):
- MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center — http://www.mdanderson.org